CLINICAL TRIAL: NCT00226135
Title: Lamotrigine Versus Lithium in Subjects With Bipolar Affective Disorders - a Randomised Study of Prophylactic Effect
Brief Title: Prophylactic Effect of Lamotrigine Compared With Lithium in Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Stanley Medical Research Institute (Other); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2612-1400; 98-rc-316
Record Dates: First submitted 2005-09-23; First posted 2005-09-26 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Treatment; Long-term; Lithium; Lamotrigine; Randomised Clinical Trial
MeSH Terms: conditions — Bipolar Disorder | interventions — Lithium; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lithium or lamotrigine

SUMMARY:
The purpose of this study is to compare lamotrigine with lithium in the long term treatment of bipolar disorder in terms of new episode preventive potentials.

DETAILED DESCRIPTION:
Bipolar disorder is a recurrent lifelong illness. Lithium is still the drug of first choice in the prophylactic treatment. However, lithium's side effects are considerable. Thus the interest in developing alternatives to lithium has increased, and various antiepileptic drugs have been studied. Among these, lamotrigine, which generally is well tolerated, has been evaluated in industry generated trials. However, for various reasons, the generalisability of the results from these studies is limited. Also the follow-up time is limited. This study is a pragmatic effectiveness study, overcoming some of these limitations, and comparing lamotrigine with that of lithium in terms of their potentials for preventing new episodes in patients with bipolar disorder.

ELIGIBILITY:
Inclusion criteria:

1. Age above 18
2. Inclusion is preceded by an affective episode requiring hospitalisation or outpatient drug treatment (index episode) which can be a manic episode (ICD-10 research criteria), a depressive episode of at least moderate degree (ICD-10 research criteria) or a mixed manic state (manic episode with at least additional three ICD-10 depressive symptoms except for difficulties with concentration or thinking, agitation or dyssomnia). The episode can be with or without psychotic symptoms including Schneiderian first-rank symptoms or bizarre delusions as long as the psychotic symptoms do not occur outside the affective episode.
3. No more than 12 months may pass between the onset of the index episode (or admission if that is the case)and date of randomisation (in order to ensure a current risk of relapse as well as reliable psychopathological information).
4. Besides the index episode, at least one previous episode must have occurred within the last five years which meets the criteria mentioned in point number two above. This episode may not necessarily have led to hospitalisation. Two episodes are separated by at least two months without significant symptoms or change in polarity (depression to mania/mixed mania or vice versa).
5. At least one manic episode (or mixed manic episode) within the last 5 years.

Exclusion criteria:

1. Contraindications to the protocol drugs.
2. Severe somatic disease, e.g. epilepsy, which may interfere with study treatment or effect evaluation.
3. Pregnancy (or risk of pregnancy).
4. Subject has prior to randomization received prophylactic treatment with lithium or lamotrigine conducted adequately in the sense of sufficient time and dose and ensuring compliance, and experienced a definite lack of prophylactic effect
5. An ICD-10 diagnosis of abuse within the last year with a subsequent risk of protocol violation. Therefore, subjects with a secondary abuse can often be included in the study.
6. Anticipated protocol violation for other reasons.
7. No written informed consent from the subject can be obtained.
8. The subject has previously been randomised in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2001-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Time to a new mood episode after having succeeded the first 6 month of treatment and reached monotherapy with study drug at that point. New episode defined as symptoms requiring treatment or admission (or suicide).

SECONDARY OUTCOMES:
1: number of patients (ITT population)that completed first 6 months and achieved monotherapy at that time.
2: Number of patients with reported AE (type specified)
3: Number of patients with an endpoint other than censoring (among populations under observation for ½ year, 1 year, 1½ years, 2 years, and 2½ years)
4:The primary end point but selected to patients under observations for 1½ and 2½ years
5: Number of endpoint (other than censoring)among patients reaching 6 months and monotherapy at that time, per person-time(testing for inter-group balance with respect to background variables)

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus W Licht, MD, PhD, Principal Investigator — Aarhus University Psychiatric Hospital, Risskov, Denmark
Locations (1):
- Aarhus University Psychiatric Hospital, Risskov, Risskov, Denmark

REFERENCES:
- [Derived] Hashimoto Y, Kotake K, Watanabe N, Fujiwara T, Sakamoto S. Lamotrigine in the maintenance treatment of bipolar disorder. Cochrane Database Syst Rev. 2021 Sep 15;9(9):CD013575. doi: 10.1002/14651858.CD013575.pub2. PMID 34523118